CLINICAL TRIAL: NCT01394432
Title: Endocardial Mesenchymal Stem Cells Implantation in Patients After Acute Myocardial Infarction
Brief Title: "ESTIMATION Study" for Endocardial Mesenchymal Stem Cells Implantation in Patients After Acute Myocardial Infarction
Acronym: ESTIMATION
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RBI-1749; RU8HM86-54N (Other: State Research Institute of Circulation Pathology)
Record Dates: First submitted 2011-07-08; First posted 2011-07-14 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Acute Myocardial Infarction; Heart Failure
Keywords: Endocardial Stem Cells Injection; Percutaneous Coronary Intervention
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (PCI+SC implantation) (Active Comparator): Endocardial Stem cells implantation with Noga system
  Interventions: Procedure: PCI and Stem Cells or Placebo injections
- Group 2 (PCI+Placebo) (Placebo Comparator): Placebo
  Interventions: Procedure: PCI and Stem Cells or Placebo injections

INTERVENTIONS:
Procedure: PCI and Stem Cells or Placebo injections — Conventional percutaneous coronary intervention after acute myocardial infarction. Harvest of bone marrow from iliac crest. Mesenchymal autologous stem cells preparation (7-10 days after PCI). LV mapping with Noga system (7-10 days after PCI). Randomization 1:1. Stem Cells or placebo implantation.

SUMMARY:
The investigators hypothesised that endocardial stem cells implantation following after percutaneous coronary intervention (PCI) could reduce the scar formation and increase reverse remodeling in patients with primary acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute Q-wave myocardial infarction after thrombolitic therapy during 6-36 hours from the onsent of signs
* Oclusion or significant stenosis of infarct-related left anterior descending artery (LAD)
* Left ventricle ejection fraction (LVEF) < 50% measured by Echo

Exclusion Criteria:

* Thrombolysis of pyrrolase or streptokinase
* Surgical unsignificant stenosis of LAD
* Indications for CABG
* Cardiogenic shock
* Uncontrolled hypertension
* Thrombocytopenia
* Ongoing bleeding
* Anemia < 100 g/l
* Oncology
* Patients, who required anticoagulation therapy at the time of inclusion
* Obesity, BMI>40
* Severe comorbidities
* Unwillingness to participate

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-11 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Reduction in left ventricle systolic volume on 15% mesured by MRI | 12 months

SECONDARY OUTCOMES:
All-cause death | 12 months
number of patients with thromboembolic events | 12 months
  comparison the number of patients with thromboembolic events between two groups
number of heart failure hospitalizations | 12 months
Distance during 6-minute walking test | 12 months
number of patients with life-threatening arrhythmias | 12 months
BNP level | 12 months
SPECT and Echo data | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny A Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia